CLINICAL TRIAL: NCT04008355
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess Tolerability, Safety, Pharmacokinetics and Effect of AZP2006 on Cerebrospinal Fluid Biomarkers in 36 Patients With Progressive Supranuclear Palsy
Brief Title: A Study to Assess Tolerability, Safety, Pharmacokinetics and Effect of AZP2006 in Patients With PSP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlzProtect SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AZP2006C04
Record Dates: First submitted 2019-06-18; First posted 2019-07-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 60mg/day/84 days (Experimental): Patients randomized in this arm will receive 60 mg of study investigational drug AZP2006 once daily during 84 days.
  Interventions: Drug: AZP2006 oral solution
- 80mg/day/10 days followed by 50mg/day/74 days (Experimental): Patients randomized in this arm will receive 80 mg of study investigational drug AZP2006 once daily during 10 days followed by 50 mg of study investigational drug AZP2006 once daily during the next 74 days.
  Interventions: Drug: AZP2006 oral solution
- Placebo/84 days (Placebo Comparator): Patients randomized in this arm will receive placebo solution once daily during 84 days.
  Interventions: Drug: Placebo oral solution

INTERVENTIONS:
Drug: AZP2006 oral solution — Once daily intake in the morning
  Arms: 60mg/day/84 days; 80mg/day/10 days followed by 50mg/day/74 days
Drug: Placebo oral solution — Once daily intake in the morning
  Arms: Placebo/84 days

SUMMARY:
A phase 2 study to assess tolerability, safety, pharmacokinetics and effect of AZP2006 at different doses versus placebo on cerebrospinal fluid biomarkers in 36 patients with progressive supranuclear palsy. The patient study duration is 29 weeks including a washout period.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, parallel group study comparing 2 doses of AZP2006 (60 mg Once daily [QD] during the 12-week treatment period or 80 mg for 10 days followed by 50 mg QD) with placebo in 36 men and women aged ≥40 years and ≤80 years and diagnosed with probable or possible PSP according to Movement Disorder Society PSP (MDS-PSP) criteria.

Patients were assessed for eligibility at baseline. Eligible patients were randomized on

Day -1 in a 1:1:1 ratio into one of the following 3 study intervention groups based on a randomization scheme with blocks stratified by center using an interactive web response system (IWRS):

1. 60 mg AZP2006/day during the 12-week treatment period;
2. 80 mg AZP2006/day for 10 days followed by 50 mg AZP2006/day;
3. Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with probable or possible PSP
* Patients must be stable with their medication for at least 30 days prior to the inclusion visit.

Exclusion Criteria:

* Any history of clinically significant head trauma or cerebrovascular disease or recent history of substance abuse or alcohol abuse and deemed to be clinically significant by the Investigator.
* History of deep brain stimulator (DBS) surgery other than sham surgery for DBS clinical study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients who prematurely discontinue from the study due to adverse events (AEs) | From Day 1 to Day 180
  Incidence in pourcentage of treatment-emergent adverse events observed directly by investigator and adverse event spontaneously reported by the patient using concise medical terminology
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the Cmax of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the tmax of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the kel of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the Clast of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the AUC 0-10 of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the AUC 0-24 of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the AUC 0-t of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the t1/2 of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the tlast of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the %AUCextra of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the CL/F of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the Vd/F of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks
The pharmacokinetics of AZP2006 (12-week treatment period) in plasma, blood, and CSF | From Day 1 of Day 84 (12 weeks)
  To determine the Ctrough of AZP2006 in plasma, blood, and CSF after single and multiple dose administration, once daily for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Verwaerde, PhD, Study Director — AlzProtect SAS
Locations (3):
- France (3):
  - Hôpital Salengro, Lille, Hauts-de-France
  - Hôpital de la Fondation Adolphe de Rothschild, Paris
  - Hôpitaux Universitaires Pitié Salpêtrière - Charles Foix, Paris, Île-de-France Region